CLINICAL TRIAL: NCT02338154
Title: Assessing Standard oF Care and Clinical Outcomes UsiNg the EDWARDS INTUITY VAlve SysTem in a European multI-center, Active, pOst-market surveillaNce Study.
Brief Title: EDWARDS INTUITY Valve System FOUNDATION Study
Acronym: FOUNDATION
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-13
Record Dates: First submitted 2014-11-19; First posted 2015-01-14 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Aortic Valve Disease; Aortic Stenosis; Rapid Deployment Valves
Keywords: Aortic Valve Replacement; Aortic Stenosis; EDWARDS INTUITY
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this active post-market surveillance study is to confirm the safety and effectiveness of the EDWARDS INTUITY Valve System in the study population.

The objective is to evaluate cardiac performance characteristics and adverse events rates associated with the EDWARDS INTUITY Valve in patients undergoing AVR. The AVR surgical approach is either full or partial sternotomy or a right anterior thoracotomy.

DETAILED DESCRIPTION:
Aortic valve replacement with mechanical or biological heart valves is the treatment of choice for aortic valve stenosis. Over the past several years, life expectancy has increased in industrial nations, but this has been accompanied by a rising rate of elderly patients with multiple illnesses.

Aortic stenosis remains the most common cause of adult valvular heart disease, the prevalence increasing with age. Average survival of patients treated conservatively has historically been reported as 2-5 years from the onset of symptoms. More recent studies have confirmed the dismal prognosis of severe aortic stenosis. Advanced age, reduced left ventricular ejection fraction, congestive heart failure and renal insufficiency appear to be independent predictors of reduced survival. Asymptomatic patients with very severe aortic stenosis also share a poor prognosis with a high event rate and a risk of rapid functional deterioration. Early surgery offers a therapeutic option to improve clinical outcomes via decreasing cardiac mortality and improving symptoms.

Bioprostheses offer several advantages over mechanical bioprostheses, the most important being freedom from anticoagulation with a low rate of thromboembolic accidents.

In response to clinical need and in support of advances in minimally invasive surgical approaches to conventional AVR, Edwards Lifesciences developed the EDWARDS INTUITY Valve System to achieve clinical benefits by reducing cardiopulmonary bypass and cross clamp times, while facilitating a less invasive approach to aortic valve replacement.

The system includes the EDWARDS INTUITY Valve System, Model 8300A and the EDWARDS INTUITY Delivery System, Model 8300D; the valve is based on prior heart valve designs which have a long history of safety and effectiveness and have incorporated additional features designed to improve patient outcomes and safety.

With only 3 guiding sutures and secure balloon expandable frame, the EDWARDS INTUITY Valve system is well suited for smaller incisions and tight access, with an emphasis on procedural efficiency within existing operating suite of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject presents with aortic stenosis or stenosis-based insufficiency of an aortic valve requiring a planned replacement of the native aortic valve or previously implanted aortic prosthesis.
3. Subject has signed and dated the investigation informed consent forms prior to study-specific procedures are performed.
4. Subject is geographically stable and agrees to attend follow-up assessments as specified in the protocol and informed consent.

Exclusion Criteria:

1. History of active endocarditis within three months of scheduled surgery
2. Subject is diagnosed with pure aortic insufficiency
3. Aneurysm of the aortic root and/or ascending aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects, age 18 or older, that have been diagnosed with aortic stenosis or stenosis-based insufficiency and are scheduled to undergo surgical aortic valve replacement are eligible for participation in this study. Study subjects shall be drawn from the general patient populations served by each investigational center. Candidates for this study must meet all of the following inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Glauber, MD, Principal Investigator — Organizational Affiliation: OSPEDALE "G. PASQUINUCCI" CREAS IFC-CNR; Prof.Christopher Young, MD FRCS, Principal Investigator — Guy's & St Thomas' Hospital
Locations (27):
- Austria (3):
  - Salzburger Universitätsklinikum, Salzburg
  - Landesklinikum - St. Pölten, Sankt Pölten
  - Klinisshe Abteiluing Für Herz-thoraxchirurgie, Vienna
- Aarhus Universitetshospital Skejby, Aarhus N, Denmark
- France (4):
  - CHU Bocage Central Dijon, Dijon
  - Hôpital Saint Joseph - Marseille, Marseille
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Cardiologique du Nord St Denis, Saint-Denis
- Germany (3):
  - Herz- und Gefäß-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale
  - Westdeutsches Herzcentrum Uniklinik Essen, Essen
  - Klinikum Nürnberg Süd, Nürenberg
- Italy (7):
  - Clinica Santa Maria, Bari
  - S. Anna Hospital, Catanzaro
  - G. Pasquinucci Heart Hospital - "G.Monasterio" Foundation, Massa
  - Centro Cardiologico Monzino, Milan
  - Ospedale Niguarda Ca' Granda, Milan
  - Università Cattolica del Sacro Cuore Policlinico, Roma
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine
- Catharina Hospital Eindhoven, Eindhoven, Netherlands
- Spain (3):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Cruces Barakaldo, Barakaldo
  - Hospital Clínico San Carlos, Madrid
- Switzerland (3):
  - Universitätsklinik Für Herz und Gefässchirurgie, Bern
  - Cardiocentro Ticino, Lugano
  - Universität Zurich, Zurich
- United Kingdom (2):
  - St Thomas' Hospital, London
  - King's College Hospital, London

REFERENCES:
- [Result] Young C, Laufer G, Kocher A, Solinas M, Alamanni F, Polvani G, Podesser BK, Aramendi JI, Arribas J, Bouchot O, Livi U, Massetti M, Terp K, Giot C, Glauber M. One-year outcomes after rapid-deployment aortic valve replacement. J Thorac Cardiovasc Surg. 2018 Feb;155(2):575-585. doi: 10.1016/j.jtcvs.2017.09.133. Epub 2017 Oct 31. PMID 29415382

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 516 Subjects were enrolled in this study, for which data is available.
Groups:
- EDWARDS INTUITY Aortic Valve: Aortic valve replacement therapy Heart Valve Surgery: The system includes the EDWARDS INTUITY Valve System, Model 8300A and the EDWARDS INTUITY Delivery System, Model 8300D
Period: Overall Study
Arm/Group | EDWARDS INTUITY Aortic Valve
Started | 516
Enrolled Cohort (Intent to Treat) | 516
INTUITY (Study Valve Cohort) | 493
Completed | 373
Not Completed | 143
Not completed — Death | 46
Not completed — Valve Implant Failure | 17
Not completed — Valve Explant | 11
Not completed — Withdrawal by Subject or by Investigator | 10
Not completed — Lost to Follow-up | 8
Not completed — Other Reason | 3
Not completed — Patients Without Exit Form | 47
Not completed — Missing Exit Reason on Exit Form | 1

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Cohort: Subjects were considered enrolled into the clinical study when he/she signed the informed consent, met all the study eligibility criteria, and after the surgeon placed the first guiding suture on the bioprosthesis.
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 516
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed is the number of patients with available data for the given parameter.
  years
    number analyzed (Participants) | 515
    (all) | 75.5 (6.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 223
  Male | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed is the number of patients with available data for the given parameter.
  Participants
    number analyzed (Participants) | 458
    Hispanic or Latino | 218
    Not Hispanic or Latino | 240
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed is the number of patients with available data for the given parameter.
  Participants
    number analyzed (Participants) | 458
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 456
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject's Average Time Spent on Cardiopulmonary Cross Clamp
Description: Cardiopulmonary cross clamp time is the amount of time that the patient's aorta (blood vessel) is clamped by a surgical instrument used in cardiac surgery. This allows the normal blood flow to be sent to an artificial heart and lung machine to keep it at a constant temperature and oxygen level.
Time Frame: At time of surgery; an average of 1 hour
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- INTUITY (Study Valve Cohort): The study valve cohort consists of all patients that left the operating room with the study valve in place.
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 476
minutes | 59.7 (24.0)

2. Other Pre Specified Outcome: Subject's Average Time Spent on Cardiopulmonary Bypass
Description: Cardiopulmonary bypass time is the amount of time that the patient's blood circulates through an artificial heart and lung machine during cardiac surgery.
Time Frame: At time of surgery; an average of 1.5 hours
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 474
minutes | 85.9 (33.0)

3. Other Pre Specified Outcome: Subject's Average Skin-to-skin Time
Description: The time from start of skin incision to end of skin closure.
Time Frame: At time of surgery; an average of 3.5 hours
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 478
Minutes | 199.3 (69.8)

4. Other Pre Specified Outcome: Subject's Device Technical Success
Description: Device technical success is defined as the successful delivery and deployment of the aortic trial heart valve with the subject leaving the operating room (OR) with valve in place.
Time Frame: At time of surgery
Population: The outcome is reported for subjects where data is available.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Cohort: Subject were considered enrolled into the clinical study when he/she signed the informed consent, met all the study eligibility criteria, and after the surgeon placed the first guiding suture on the bioprosthesis.
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 516
Participants | 493

5. Other Pre Specified Outcome: Subject's Average Health Care Utilization
Description: The average amount of time the subjects spent in the intensive care unit and the average total length of hospital stay after their heart valve replacement procedure.
Time Frame: Day of surgical procedure through discharge from the ICU and hospital, an average of 3 days and 11 days respectively.
Population: The outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 516
Days
  ICU Length of Stay: number analyzed (Participants) | 492
  ICU Length of Stay | 2.8 (3.9)
  Hospital Length of Stay: number analyzed (Participants) | 507
  Hospital Length of Stay | 11.2 (18.4)

6. Other Pre Specified Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: 30 days, 3 months, 1 year, 2 years
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 493
Participants
  30 Days: number analyzed (Participants) | 418
  30 Days: Improved | 272
  30 Days: Same | 129
  30 Days: Worsened | 17
  3 Months: number analyzed (Participants) | 433
  3 Months: Improved | 326
  3 Months: Same | 99
  3 Months: Worsened | 8
  1 Year: number analyzed (Participants) | 364
  1 Year: Improved | 293
  1 Year: Same | 63
  1 Year: Worsened | 8
  2 Year: number analyzed (Participants) | 350
  2 Year: Improved | 255
  2 Year: Same | 80
  2 Year: Worsened | 15

7. Other Pre Specified Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline, 3 months
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 493
units on a scale
  Baseline: number analyzed (Participants) | 172
  Baseline | 0.818 (0.137)
  3 Months: number analyzed (Participants) | 162
  3 Months | 0.864 (0.149)
  Change from Baseline to 3 Months: number analyzed (Participants) | 157
  Change from Baseline to 3 Months | 0.040 (0.131)

8. Other Pre Specified Outcome: Subject's Average Mean Gradient Measurements
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Baseline, discharge, 3 months, and 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- INTUITY (Study Valve Cohort) - 19mm; INTUITY (Study Valve Cohort) - 21mm; INTUITY (Study Valve Cohort) - 23mm; INTUITY (Study Valve Cohort) - 25mm; INTUITY (Study Valve Cohort) - 27mm; INTUITY (Study Valve Cohort) - Overall: The study valve cohort consists of all patients that left the operating room with the study valve in place.
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
mmHg
  Baseline: number analyzed (Participants) | 67 | 117 | 141 | 85 | 25 | 435
  Baseline | 51.22 (21.24) | 49.11 (16.81) | 47.51 (16.70) | 44.36 (13.33) | 44.83 (14.79) | 47.74 (16.90)
  Discharge: number analyzed (Participants) | 69 | 126 | 139 | 84 | 27 | 445
  Discharge | 15.83 (8.35) | 11.74 (6.42) | 10.69 (5.98) | 10.69 (7.65) | 7.77 (2.96) | 11.61 (7.00)
  3 months: number analyzed (Participants) | 62 | 107 | 133 | 82 | 26 | 410
  3 months | 14.58 (8.26) | 10.96 (6.01) | 9.73 (5.98) | 8.34 (4.68) | 7.38 (2.80) | 10.36 (6.34)
  1 Year: number analyzed (Participants) | 50 | 91 | 110 | 67 | 28 | 346
  1 Year | 13.16 (6.90) | 10.14 (4.28) | 8.96 (3.72) | 8.45 (3.03) | 7.25 (3.13) | 9.64 (4.60)

9. Other Pre Specified Outcome: Subject's Average Peak Gradients (mmHg) Measurements Over Time
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: Baseline, discharge, 3 months, and 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
mmHg
  Baseline: number analyzed (Participants) | 67 | 119 | 144 | 86 | 25 | 441
  Baseline | 83.75 (33.17) | 78.92 (28.21) | 77.08 (25.15) | 73.11 (20.92) | 72.51 (21.22) | 77.56 (26.55)
  Discharge: number analyzed (Participants) | 69 | 126 | 141 | 85 | 28 | 449
  Discharge | 29.42 (12.83) | 21.88 (10.53) | 20.29 (9.75) | 19.78 (12.28) | 14.00 (5.63) | 21.65 (11.40)
  3 Months: number analyzed (Participants) | 62 | 109 | 134 | 82 | 26 | 413
  3 Months | 27.46 (13.64) | 21.12 (10.32) | 19.48 (11.90) | 16.52 (7.82) | 14.00 (4.96) | 20.18 (11.32)
  1 Year: number analyzed (Participants) | 50 | 93 | 109 | 69 | 28 | 349
  1 Year | 23.88 (8.57) | 18.29 (7.17) | 16.97 (6.77) | 15.40 (4.94) | 13.29 (5.37) | 17.70 (7.31)

10. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Measurements
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Baseline, discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: Centimeters squared
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
Centimeters squared
  Baseline: number analyzed (Participants) | 59 | 108 | 132 | 78 | 20 | 397
  Baseline | 0.62 (0.16) | 0.71 (0.29) | 0.75 (0.34) | 0.74 (0.26) | 0.81 (0.25) | 0.72 (0.29)
  Discharge: number analyzed (Participants) | 58 | 99 | 122 | 68 | 20 | 367
  Discharge | 1.17 (0.41) | 1.66 (0.53) | 2.00 (0.64) | 2.18 (0.70) | 2.83 (0.90) | 1.86 (0.73)
  3 Months: number analyzed (Participants) | 56 | 99 | 119 | 77 | 24 | 375
  3 Months | 1.14 (0.39) | 1.59 (0.52) | 1.86 (0.62) | 2.10 (0.59) | 2.54 (0.77) | 1.77 (0.67)
  1 Year: number analyzed (Participants) | 45 | 83 | 98 | 60 | 26 | 312
  1 Year | 1.28 (0.33) | 1.61 (0.43) | 1.97 (0.42) | 2.23 (0.65) | 2.64 (0.73) | 1.88 (0.63)

11. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurements
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: Baseline, Discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Groups:
- INUTITY (Study Valve Cohort) - 19mm; INTUITY (Study Valve Cohort) - 21mm; INTUITY (Study Valve Cohort) - 23mm; INTUITY (Study Valve Cohort) - 25mm; INTUITY (Study Valve Cohort) - 27mm; INTUITY (Study Valve Cohort) - Overall: The study valve cohort consists of all patients that left the operating room with the study valve in place.
Arm/Group | INUTITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
centimeters squared/meters squared
  Baseline: number analyzed (Participants) | 59 | 108 | 129 | 78 | 20 | 394
  Baseline | 0.37 (0.10) | 0.41 (0.18) | 0.40 (0.17) | 0.37 (0.14) | 0.40 (0.12) | 0.39 (0.16)
  Discharge: number analyzed (Participants) | 49 | 79 | 94 | 54 | 18 | 294
  Discharge | 0.69 (0.26) | 0.92 (0.31) | 1.05 (0.34) | 1.15 (0.35) | 1.40 (0.50) | 0.99 (0.38)
  3 Months: number analyzed (Participants) | 48 | 87 | 89 | 58 | 20 | 302
  3 Months | 0.69 (0.24) | 0.91 (0.31) | 0.99 (0.40) | 1.09 (0.34) | 1.23 (0.42) | 0.96 (0.37)
  1 Year: number analyzed (Participants) | 41 | 79 | 94 | 52 | 21 | 287
  1 Year | 0.76 (0.21) | 0.92 (0.26) | 1.06 (0.22) | 1.13 (0.33) | 1.30 (0.48) | 1.01 (0.31)

12. Other Pre Specified Outcome: Subject's Average Performance Index Measurements
Description: Performance index is defined as the subject's effective orifice area (the cross-sectional area of the blood flow downstream of the aortic valve) divided by the subject's native orifice area. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/cm^2
Arm/Group | INUTITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
cm^2/cm^2
  Discharge: number analyzed (Participants) | 54 | 97 | 103 | 69 | 22 | 345
  Discharge | 0.44 (0.12) | 0.49 (0.13) | 0.53 (0.14) | 0.49 (0.12) | 0.56 (0.12) | 0.50 (0.13)
  3 Months: number analyzed (Participants) | 46 | 87 | 104 | 72 | 23 | 332
  3 Months | 0.44 (0.12) | 0.50 (0.12) | 0.55 (0.13) | 0.52 (0.13) | 0.57 (0.13) | 0.52 (0.13)
  1 Year: number analyzed (Participants) | 45 | 75 | 89 | 56 | 22 | 287
  1 Year | 0.48 (0.12) | 0.51 (0.14) | 0.55 (0.12) | 0.53 (0.13) | 0.58 (0.13) | 0.53 (0.13)

13. Other Pre Specified Outcome: Subject's Average Left Ventricular Ejection Fraction (LVEF)
Description: Ejection fraction is a measurement of the percentage of blood leaving your heart each time it contracts. Ejection fraction is evaluated by echocardiography over time. A normal left ventricular ejection fraction (LVEF) ranges from 55% to 70%.
Time Frame: Baseline, discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Mean (Standard Deviation); unit: Percentage of blood
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
Percentage of blood
  Baseline: number analyzed (Participants) | 66 | 112 | 134 | 83 | 23 | 418
  Baseline | 66.71 (9.85) | 65.87 (11.89) | 64.56 (11.73) | 60.57 (12.85) | 62.96 (9.29) | 64.37 (11.75)
  Discharge: number analyzed (Participants) | 66 | 113 | 132 | 74 | 25 | 410
  Discharge | 66.05 (11.40) | 64.16 (11.63) | 65.87 (10.70) | 60.45 (12.57) | 61.12 (13.36) | 64.16 (11.73)
  3 Months: number analyzed (Participants) | 57 | 105 | 128 | 81 | 26 | 397
  3 Months | 64.58 (6.96) | 66.26 (9.88) | 65.20 (9.51) | 62.36 (11.29) | 63.08 (10.24) | 64.67 (9.79)
  1 Year: number analyzed (Participants) | 40 | 76 | 93 | 62 | 22 | 293
  1 Year | 64.28 (8.12) | 64.64 (8.23) | 64.65 (8.98) | 63.30 (7.75) | 63.64 (9.35) | 64.23 (8.41)

14. Other Pre Specified Outcome: Subject's Amount of Aortic Valvular Regurgitation Over Time.
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: Discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
Participants
  Discharge: number analyzed (Participants) | 68 | 118 | 134 | 78 | 26 | 429
  Discharge: 0 None | 34 | 69 | 83 | 52 | 19 | 260
  Discharge: +1 Trivial/Trace | 29 | 39 | 42 | 22 | 6 | 140
  Discharge: +2 Mild | 5 | 9 | 9 | 4 | 1 | 28
  Discharge: +3 Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Discharge: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  3 Months: number analyzed (Participants) | 61 | 116 | 137 | 83 | 30 | 430
  3 Months: 0 None | 25 | 67 | 80 | 55 | 21 | 249
  3 Months: +1 Trivial/Trace | 28 | 39 | 43 | 24 | 8 | 144
  3 Months: +2 Mild | 7 | 7 | 9 | 4 | 1 | 28
  3 Months: +3 Moderate | 1 | 2 | 5 | 0 | 0 | 8
  3 Months: +4 Severe | 0 | 1 | 0 | 0 | 0 | 1
  1 Year: number analyzed (Participants) | 50 | 93 | 116 | 69 | 28 | 358
  1 Year: 0 None | 29 | 60 | 78 | 49 | 18 | 236
  1 Year: +1 Trivial/Trace | 15 | 23 | 21 | 17 | 9 | 85
  1 Year: +2 Mild | 5 | 9 | 12 | 3 | 1 | 30
  1 Year: +3 Moderate | 1 | 1 | 3 | 0 | 0 | 5
  1 Year: +4 Severe | 0 | 0 | 2 | 0 | 0 | 2

15. Other Pre Specified Outcome: Subject's Amount of Paravalvular Leak Over Time.
Description: Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing. Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
Participants
  Discharge: number analyzed (Participants) | 67 | 118 | 137 | 79 | 24 | 430
  Discharge: 0 None | 59 | 99 | 105 | 69 | 22 | 358
  Discharge: +1 Trivial/Trace | 4 | 18 | 25 | 6 | 1 | 55
  Discharge: +2 Mild | 4 | 1 | 6 | 4 | 1 | 16
  Discharge: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Discharge: +4 Severe | 0 | 0 | 1 | 0 | 0 | 1
  3 Months: number analyzed (Participants) | 60 | 110 | 130 | 82 | 28 | 413
  3 Months: 0 None | 52 | 84 | 96 | 67 | 22 | 324
  3 Months: +1 Trivial/Trace | 5 | 20 | 22 | 11 | 5 | 63
  3 Months: +2 Mild | 3 | 6 | 12 | 4 | 1 | 26
  3 Months: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  3 Months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: number analyzed (Participants) | 43 | 83 | 96 | 65 | 24 | 313
  1 Year: 0 None | 32 | 64 | 65 | 56 | 20 | 238
  1 Year: +1 Trivial/Trace | 9 | 17 | 16 | 6 | 4 | 53
  1 Year: +2 Mild | 1 | 2 | 14 | 3 | 0 | 20
  1 Year: +3 Moderate | 1 | 0 | 1 | 0 | 0 | 2
  1 Year: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Subject's Average Cardiac Output Over Time
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: Discharge, 3 months, 1 year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
liters per minute
  Discharge: number analyzed (Participants) | 54 | 94 | 106 | 67 | 20 | 341
  Discharge | 4.14 (1.39) | 4.24 (1.31) | 4.60 (1.33) | 4.74 (1.48) | 5.09 (1.82) | 4.49 (1.42)
  3 Months: number analyzed (Participants) | 47 | 88 | 104 | 74 | 20 | 333
  3 Months | 3.85 (1.40) | 4.36 (1.15) | 4.29 (1.12) | 4.16 (1.19) | 5.08 (1.57) | 4.26 (1.23)
  1 Year: number analyzed (Participants) | 44 | 75 | 89 | 56 | 21 | 285
  1 Year | 3.86 (1.28) | 4.26 (1.11) | 4.61 (1.30) | 4.61 (1.30) | 5.90 (1.76) | 4.50 (1.37)

17. Other Pre Specified Outcome: Subject's Average Cardiac Output Index
Description: A hemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA).
Time Frame: Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
L/min/m2
  Discharge: number analyzed (Participants) | 45 | 73 | 79 | 53 | 18 | 268
  Discharge | 2.45 (0.89) | 2.40 (0.79) | 2.44 (0.75) | 2.54 (0.72) | 2.45 (0.77) | 2.45 (0.78)
  3 Months: number analyzed (Participants) | 39 | 77 | 77 | 53 | 19 | 265
  3 Months | 2.40 (0.88) | 2.54 (0.67) | 2.33 (0.62) | 2.21 (0.65) | 2.61 (1.00) | 2.40 (0.72)
  1 Year: number analyzed (Participants) | 40 | 72 | 85 | 48 | 16 | 261
  1 Year | 2.32 (0.81) | 2.47 (0.68) | 2.49 (0.71) | 2.32 (0.65) | 2.88 (1.09) | 2.45 (0.74)

18. Other Pre Specified Outcome: Subject's Average Left Ventricular End-Diastolic Dimension
Description: The measurement of the heart's left ventricle at end diastole.
Time Frame: Baseline, Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
centimeters
  Baseline: number analyzed (Participants) | 53 | 106 | 121 | 74 | 17 | 371
  Baseline | 4.05 (0.58) | 4.30 (0.74) | 4.38 (0.63) | 4.76 (0.72) | 4.92 (0.67) | 4.41 (0.72)
  Discharge: number analyzed (Participants) | 40 | 80 | 98 | 56 | 19 | 293
  Discharge | 3.92 (0.67) | 4.09 (0.68) | 4.35 (0.65) | 4.51 (0.73) | 4.67 (1.30) | 4.27 (0.76)
  3 Months: number analyzed (Participants) | 43 | 86 | 102 | 71 | 21 | 323
  3 Months | 3.93 (0.59) | 4.17 (0.59) | 4.25 (0.62) | 4.55 (0.68) | 4.88 (0.79) | 4.29 (0.67)
  1 Year: number analyzed (Participants) | 38 | 62 | 75 | 49 | 21 | 245
  1 Year | 3.98 (0.64) | 4.08 (0.71) | 4.43 (0.54) | 4.47 (0.72) | 4.72 (0.64) | 4.30 (0.68)

19. Other Pre Specified Outcome: Subject's Average Left Ventricular End-Systolic Dimension
Description: The measurement of the heart's left ventricle at end systole.
Time Frame: Baseline, Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | INTUITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
centimeters
  Baseline: number analyzed (Participants) | 53 | 104 | 118 | 73 | 17 | 365
  Baseline | 2.63 (0.60) | 2.80 (0.75) | 2.99 (0.72) | 3.29 (0.91) | 3.36 (0.82) | 2.96 (0.79)
  Discharge: number analyzed (Participants) | 40 | 80 | 97 | 54 | 19 | 290
  Discharge | 2.60 (0.65) | 2.80 (0.73) | 2.97 (0.69) | 3.07 (0.70) | 3.32 (0.84) | 2.92 (0.72)
  3 Months: number analyzed (Participants) | 43 | 86 | 102 | 71 | 21 | 323
  3 Months | 2.53 (0.56) | 2.70 (0.62) | 2.81 (0.56) | 3.02 (0.67) | 3.31 (0.75) | 2.82 (0.64)
  1 Year: number analyzed (Participants) | 38 | 62 | 74 | 49 | 20 | 243
  1 Year | 2.63 (0.61) | 2.69 (0.69) | 2.90 (0.54) | 2.91 (0.68) | 3.06 (0.68) | 2.82 (0.64)

20. Other Pre Specified Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Left Ventricular end-diastolic volume (LVEDV) is the amount of (volume) of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricle just before systole.
Time Frame: Baseline, Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | INUTITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
milliliters
  Baseline: number analyzed (Participants) | 62 | 108 | 125 | 78 | 21 | 394
  Baseline | 62.68 (23.55) | 75.17 (27.76) | 83.52 (31.17) | 101.91 (33.55) | 109.90 (41.78) | 83.00 (33.22)
  Discharge: number analyzed (Participants) | 61 | 109 | 118 | 71 | 22 | 381
  Discharge | 52.90 (20.35) | 63.26 (24.58) | 70.93 (24.61) | 82.10 (30.54) | 102.27 (39.83) | 69.74 (28.83)
  3 Months: number analyzed (Participants) | 48 | 92 | 112 | 77 | 24 | 353
  3 Months | 56.96 (24.76) | 64.89 (20.44) | 74.94 (23.96) | 91.66 (32.80) | 93.42 (31.21) | 74.78 (28.67)
  1 Year: number analyzed (Participants) | 36 | 63 | 76 | 51 | 19 | 245
  1 Year | 60.86 (21.22) | 72.46 (22.17) | 79.12 (26.37) | 85.80 (27.47) | 86.47 (31.99) | 76.69 (26.49)

21. Other Pre Specified Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Left Ventricular end-systolic volume (LVESV) is the amount of (volume) of blood in the left ventricle at the end of the heart's contraction, or systole, and the beginning of filling, or diastole.
Time Frame: Baseline, Discharge, 3 Months, 1 Year
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY valve where data is available.
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | INUTITY (Study Valve Cohort) - 19mm | INTUITY (Study Valve Cohort) - 21mm | INTUITY (Study Valve Cohort) - 23mm | INTUITY (Study Valve Cohort) - 25mm | INTUITY (Study Valve Cohort) - 27mm | INTUITY (Study Valve Cohort) - Overall
Number analyzed (Participants) | 73 | 134 | 157 | 92 | 30 | 486
milliliters
  Baseline: number analyzed (Participants) | 62 | 108 | 125 | 78 | 21 | 394
  Baseline | 22 (13.47) | 27.50 (18.97) | 30.46 (19.03) | 42.36 (26.74) | 40.76 (24.75) | 31.22 (21.41)
  Discharge: number analyzed (Participants) | 61 | 109 | 118 | 71 | 22 | 381
  Discharge | 18.57 (12.38) | 23.90 (15.69) | 24.51 (13.95) | 33.27 (19.96) | 41.36 (27.97) | 25.99 (17.46)
  3 Months: number analyzed (Participants) | 48 | 92 | 112 | 77 | 24 | 353
  3 Months | 20.10 (10.93) | 22.33 (13.05) | 26.17 (14.66) | 35.77 (22.99) | 35.50 (19.66) | 27.07 (17.36)
  1 Year: number analyzed (Participants) | 36 | 63 | 76 | 51 | 19 | 245
  1 Year | 21.86 (9.28) | 26.62 (12.57) | 28.37 (14.15) | 32.00 (13.02) | 31.68 (19.08) | 27.98 (13.64)

22. Other Pre Specified Outcome: Percentage of Subjects With Early Adverse Events
Description: Number of Subjects with early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100.
Time Frame: Events occurring within 30 days of procedure
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Number; unit: Percentage of subjects
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 493
Percentage of subjects
  All cause mortality | 3.0
  Study valve-related mortality | 1.4
  Thromboembolic events | 3.9
  Study valve thrombosis | 0.2
  Bleeding event | 6.3
  All paravalvular leak | 15.0
  Major paravalvular leak (Moderate or Severe) | 1.2
  Endocarditis | 0.0
  Structural valve deterioration | 0.0
  Non-structural valve deterioration (other than PVL | 0.0
  Hemolysis | 0.4
  Reoperation | 1.2
  Explant | 0.8
  New and worsening conduction disturbance | 7.3

23. Other Pre Specified Outcome: Percentage of Late Adverse Events Divided by Late Patient Years
Description: Number of late events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 2 years post-implant
Population: This outcome is reported for subjects who received a Model 8300A Edwards INTUITY Valve where data is available.
Measure: Number; unit: Percentage of events/late patient years
Arm/Group | INTUITY (Study Valve Cohort)
Number analyzed (Participants) | 493
Percentage of events/late patient years
  All cause mortality | 3.6
  Study valve-related mortality | 1.4
  Thromboembolic events | 1.6
  Study valve thrombosis | 0.0
  Bleeding event | 0.6
  All Paravalvular Leak | 10.8
  Major paravalvular leak (Moderate or Severe) | 1.3
  Endocarditis | 0.6
  Structural valve deterioration | 0.0
  Non-structural valve deterioration (other than PVL | 0.0
  Hemolysis | 0.4
  Reoperation | 1.1
  Explant | 0.7
  New and worsening conduction disturbance | 0.0

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through two (2) years post implant
Description: Adverse event table is reported using Enrolled Cohort. Where an adverse event term below includes the word "Other", those adverse events were unable to be classified into a more specific adverse event category.
Groups:
- Enrolled Cohort: Subject's were considered enrolled into the clinical study when he/she signed the informed consent, met all the study eligibility criteria, and after the surgeon places the first guiding suture on the bioprosthesis.
Arm/Group | Enrolled Cohort
All-Cause Mortality (participants affected / at risk) | 46/516
Serious Adverse Events (participants affected / at risk) | 245/516
Other Adverse Events (participants affected / at risk) | 157/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Cohort (N=516)
Anaphylactic Reaction (General disorders) | 1 (1)
Anemia - Bleeding related - Major (Blood and lymphatic system disorders) | 2 (2)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 3 (3)
Anemia - Non-bleeding related (Blood and lymphatic system disorders) | 10 (13)
Angina, Stable (Cardiac disorders) | 1 (1)
Angina, Unstable (Cardiac disorders) | 1 (1)
Arrhythmia - AV Block - 1st degree (Cardiac disorders) | 1 (1)
Arrhythmia - AV Block - 2nd degree (Cardiac disorders) | 3 (3)
Arrhythmia - AV Block - 3rd degree (Cardiac disorders) | 25 (25)
Arrhythmia - Atrial Flutter (Cardiac disorders) | 1 (1)
Arrhythmia - Bradycardia (Cardiac disorders) | 4 (4)
Arrhythmia - Bundle Branch Block - Left (Cardiac disorders) | 3 (3)
Arrhythmia - Other (Cardiac disorders) | 5 (5)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 34 (39)
Arrhythmia - Permanent Atrial Fibrillation (Cardiac disorders) | 3 (3)
Arrhythmia - Persistant Atrial Fibrillaiton (Cardiac disorders) | 9 (12)
Arrhythmia - Tachycardia - Ventricular (Cardiac disorders) | 3 (3)
Arrhythmia - Ventricular Fibrillation (Cardiac disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Biliary (Gallbladder) (Gastrointestinal disorders) | 5 (6)
Bleeding - Cardiovascular - Major (Blood and lymphatic system disorders) | 16 (18)
Bleeding - Cardiovascular - Minor (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Gastrointestinal upper -Major (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Gastrointestinal upper -Minor (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Neurological - Major (e.g. CVA) (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Pulmonary/Respiratory - Major (e.g. hemothorax) (Blood and lymphatic system disorders) | 1 (1)
Blood Sepsis (Blood and lymphatic system disorders) | 2 (2)
Blood/ Lymphatic - Other (Blood and lymphatic system disorders) | 2 (2)
Bone Fracture/Break (Musculoskeletal and connective tissue disorders) | 8 (8)
Cancer - Newly diagnosed (General disorders) | 9 (9)
Cancer - Progression of underlying disease (General disorders) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 4 (4)
Cardiac Decompensation (Cardiac disorders) | 8 (8)
Cardiogenic Shock (Cardiac disorders) | 2 (2)
Cardiovascular - Other (Cardiac disorders) | 14 (14)
Endocarditis (Cardiac disorders) | 5 (5)
Gastrointestinal - Infection (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Genitourinary - Other (Renal and urinary disorders) | 7 (7)
Heart Failure - Acute (Cardiac disorders) | 9 (11)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 2 (2)
Hepatic complication - Other (Hepatobiliary disorders) | 1 (1)
Hypertension - Systemic (Cardiac disorders) | 4 (4)
Hypotension (Cardiac disorders) | 1 (1)
Infection /Inflammation - Other (Infections and infestations) | 5 (6)
Liver Failure - Acute (Hepatobiliary disorders) | 1 (1)
Multi-System organ failure (General disorders) | 3 (3)
Muscular Skeletal / Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 17 (18)
Myocardial Infarction (Cardiac disorders) | 1 (1)
NSD - Paravalvular Leak - +2 (General disorders) | 3 (3)
NSD - Paravalvular Leak - +3 (General disorders) | 3 (4)
NSD - Paravalvular Leak - +4 (General disorders) | 2 (2)
Nonspecific, Unknown, or Other Body System - Other complication (General disorders) | 17 (18)
Pancreatic complication (Gastrointestinal disorders) | 1 (1)
Perforation - Atrial (Cardiac disorders) | 1 (1)
Perforation - Other (Cardiac disorders) | 2 (2)
Pericardial Effusion - Major (Cardiac disorders) | 2 (2)
Pericardial Effusion - Minor (Cardiac disorders) | 1 (1)
Pericardial Tamponade - Major (Cardiac disorders) | 2 (2)
Pleural Effusion - Bilateral (Cardiac disorders) | 2 (2)
Pleural Effusion - Left (Cardiac disorders) | 4 (4)
Pleural Effusion - Right (Cardiac disorders) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychiatric - Other (Psychiatric disorders) | 1 (1)
Psychiatric Disorder (Psychiatric disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism - Bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism - Right (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Regurgitation - Aortic-Central/Transvalvular-+3 (Cardiac disorders) | 1 (1)
Regurgitation - Aortic-Central/Transvalvular-+4 (Cardiac disorders) | 1 (1)
Regurgitation - Aortic-Indeterminate-+2 (Cardiac disorders) | 1 (1)
Regurgitation - Aortic-Indeterminate-+4 (Cardiac disorders) | 1 (1)
Renal Dysfunction (Renal and urinary disorders) | 9 (9)
Renal Failure - Acute (Renal and urinary disorders) | 12 (12)
Renal Failure - Chronic (Renal and urinary disorders) | 2 (2)
Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure -COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure -Other (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Failure -Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Respiratory Failure -Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Respiratory Infection - Upper (URI) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SVD - Stent frame separation (Product Issues) | 1 (1)
Speech disorder (General disorders) | 1 (1)
Sternal Wound/Thoracic Infection (Musculoskeletal and connective tissue disorders) | 8 (10)
Suicide (Psychiatric disorders) | 1 (1)
Thromboembolic Event - Other - Central - Hemiparesis (Cardiac disorders) | 1 (1)
Thromboembolic Event - Other - Peripheral - No paresis (Cardiac disorders) | 2 (2)
Thromboembolic Event - Stroke (Cardiac disorders) | 10 (11)
Thromboembolic Event - Transient Ischemic Attack (TIA) (Cardiac disorders) | 4 (4)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 3 (5)
Valve Thrombosis - Aortic (Cardiac disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 8 (9)
NSD - Paravalvular leak with Hemolysis (General disorders) | 2 (2)
Respiratory Failure -Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Cohort (N=516)
Allergic Reaction - Medication related (General disorders) | 1 (1)
Anemia - Bleeding related - Major (Blood and lymphatic system disorders) | 1 (1)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 3 (3)
Anemia - Non-bleeding related (Blood and lymphatic system disorders) | 12 (13)
Angina, Stable (Cardiac disorders) | 1 (1)
Arrhythmia - AV Block - 1st degree (Cardiac disorders) | 2 (2)
Arrhythmia - AV Block - 3rd degree (Cardiac disorders) | 1 (1)
Arrhythmia - Bundle Branch Block - Left (Cardiac disorders) | 12 (12)
Arrhythmia - Bundle Branch Block - Right (Cardiac disorders) | 1 (1)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 46 (47)
Arrhythmia - Permanent Atrial Fibrillation (Cardiac disorders) | 4 (4)
Arrhythmia - Persistant Atrial Fibrillaiton (Cardiac disorders) | 15 (15)
Arrhythmia - Tachycardia - Ventricular (Cardiac disorders) | 1 (1)
Biliary (Gallbladder) (Gastrointestinal disorders) | 1 (1)
Bleeding - Cardiovascular - Minor (Blood and lymphatic system disorders) | 5 (5)
Bleeding - Gastrointestinal lower -Minor (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Gastrointestinal upper -Minor (Blood and lymphatic system disorders) | 3 (3)
Bleeding - Genitourinary - Minor (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Peripheral vascular - Minor (e.g. nosebleeds; hematomas) (Blood and lymphatic system disorders) | 1 (1)
Blood/ Lymphatic - Other (Blood and lymphatic system disorders) | 3 (3)
Bone Fracture/Break (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer - Newly diagnosed (General disorders) | 2 (2)
Cardiovascular - Other (Cardiac disorders) | 1 (1)
Endocrine complications (Endocrine disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 7 (7)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 2 (2)
Hepatic complication - Other (Hepatobiliary disorders) | 1 (1)
Hypertension - Systemic (Cardiac disorders) | 1 (1)
Infection /Inflammation - Other (Infections and infestations) | 3 (3)
Muscular Skeletal / Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 14 (15)
NSD - Paravalvular Leak - +2 (General disorders) | 2 (2)
NSD - Paravalvular leak with Hemolysis (General disorders) | 1 (1)
Nonspecific, Unknown, or Other Body System - Other complication (General disorders) | 3 (3)
Pericardial Effusion - Minor (Cardiac disorders) | 3 (3)
Pleural Effusion - Bilateral (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleural Effusion - Left (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychiatric - Other (Psychiatric disorders) | 6 (6)
Psychiatric Disorder (Psychiatric disorders) | 1 (1)
Pulmonary/Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Renal Dysfunction (Renal and urinary disorders) | 6 (6)
Renal Failure - Acute (Renal and urinary disorders) | 2 (2)
Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure -COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Infection - Upper (URI) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sternal Wound/Thoracic Infection (Musculoskeletal and connective tissue disorders) | 2 (2)
Thrombocytopenia - Non-Heparin Induced (Blood and lymphatic system disorders) | 5 (5)
Thromboembolic Event - Other - Peripheral - Hemiparesis (Cardiac disorders) | 1 (1)
Thromboembolic Event - Stroke (Cardiac disorders) | 1 (1)
Thromboembolic Event - Transient Ischemic Attack (TIA) (Cardiac disorders) | 3 (3)
Transient Psychotic Syndrome (Psychiatric disorders) | 5 (5)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 15 (15)
Vascular - Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)
Vision disorder (Eye disorders) | 3 (3)
Wound Infection - Other (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 30 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 60 day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.